CLINICAL TRIAL: NCT04765189
Title: Evaluation of the Efficacy of Mangoselect®, a Mangosteen Extract, and of a Formulation Containing Mangoselect®, in Subjects Suffering From Activity/Exercise-induced Knee Joint Discomfort During a 12-week Supplementation Period. A Double-blind, Randomized, Multi-arm, Parallel and Placebo-controlled Study.
Brief Title: Evaluation of Mangoselect® in Improvement of Exercise/Activity-induced Knee Joint Discomfort in Subjects Suffering From Osteoarthritis Grade I or II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MNGEFS
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Verum A (Experimental)
  Interventions: Dietary Supplement: Verum A
- Verum B (Experimental)
  Interventions: Dietary Supplement: Verum B
- Verum C (Experimental)
  Interventions: Dietary Supplement: Verum C

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo product is 100% maltodextrin. Daily dosage is 500 mg in 2 capsules.
  Arms: Placebo
Dietary Supplement: Verum A — Verum A is 200 mg of mangosteen extract. Daily dosage is 200 mg in 2 capsules.
  Arms: Verum A
Dietary Supplement: Verum B — Verum B is 400 mg of mangosteen extract. Daily dosage is 400 mg in 2 capsules.
  Arms: Verum B
Dietary Supplement: Verum C — Verum C is 200 mg mangosteen extract + 300 mg grape extract. Daily dosage is 500 mg in 2 capsules.
  Arms: Verum C

SUMMARY:
The aim of the present investigation is to evaluate the efficacy of Mangoselect®, a mangosteen extract, and of a formulation containing Mangoselect®, in subjects suffering from activity/exercise-induced knee joint pain/discomfort, during a 12-week supplementation period. Subjective discomfort improvement will be assessed with both WOMAC questionnaire and pain Visual Analogic Scale (VAS); functional joints features, quality of life, and inflammatory markers, will also be assessed. Finally, long lasting benefits will additionally be evaluated 4 weeks after the end of the supplementation period. The design of the study is double-blind, randomized, multi-arm, parallel and placebo controlled.

ELIGIBILITY:
Inclusion Criteria:

* Physically active volunteers
* BMI 22-29.9 kg/m2
* Declaring knee joint pain during and/or after activity/exercise
* Joint knee pain rated of at least 4 cm on a 10 cm VAS following activity/exercise
* Diagnosed osteoarthritis grade I or II according to Kellgren-Lawrence classification

Exclusion Criteria:

* Diagnosed inflammatory joint disorder or osteoarthritis grade III or more according to Kellgren-Lawrence classification
* Currentlu chronically taking pain killer drugs or dietary supplement or intra-articular treatment 3 months before selection
* Anemia
* Subjects with knee/joint surgery/replacement in the past 10 years
* Significant injury of the studied knee joint 12 months before selection
* Unable to carry out functional tests and/or questionnaires
* Currently participating or having participated in another clinical trial in the 3 previous months
* Pregnant women and women positive at Beta-HCG serology test
* Any condition that the investigator believes would interfere with the ability to provide inform consent, or comply with study instructions, or confound the interpretations of the study results, or put the volunteer at undue risk
* Allergy to one of the component of the supplements

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Change in knee joint pain subscale from WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) questionnaire | 12 weeks
Change in knee joint subjective pain rating using a VAS (Visual Analog Scale) 0-10 cm | 12 weeks

SECONDARY OUTCOMES:
Change in knee joint stifness subscale from WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) questionnaire | 12 weeks
Change in knee joint physical functionning subscale from WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) questionnaire | 12 weeks
Change in knee mobility assessed with ROM (Range of Motion) assessment | 12 weeks
Change in muscular strength assessed with isokinetic strength measurment | 12 weeks
Change in inflammatory status assessed with TNF-alpha plasma concentration | 12 weeks
Change in inflammatory status assessed with TNF-alpha receptor R1 plasma concentration | 12 weeks
Change in inflammatory status assessed with TNF-alpha receptor R2 plasma concentration | 12 weeks
Change in inflammatory status assessed with IL-1beta plasma concentration | 12 weeks
Change in inflammatory status assessed with IL-1beta receptor p68 plasma concentration | 12 weeks
Change in inflammatory status assessed with IL-1beta receptor p80 plasma concentration | 12 weeks
Change in quality of life assessed with SF-12 questionnaire | 12 weeks
Change in pain killer drug consumption assessed with daily diary | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Alcaraz, Principal Investigator — UCAM (Universidad Catolica San Antonio de Murcia)
Locations (1):
- UCAM (Universidad Catolica San Antonio de Murcia), Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided